CLINICAL TRIAL: NCT04169529
Title: Reveal LINQ for Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT19019
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Reveal LINQ — Insertion of Reveal LINQ device to characterize collected data from patients with COPD.

SUMMARY:
The purpose of the LINQ™ for COPD study is to characterize Reveal LINQ™ derived data from patients with COPD by assessing the relationship between changes in LINQ™ derived data with COPD exacerbation events.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is progressive and currently incurable and refers to a collection of diseases that lead to the key feature of irreversible airflow limitation and breathing related problems. Of those with COPD, 46% experienced at least one exacerbation within the previous year and 19% needed hospitalization. The financial burden of COPD is also evident, in that over $32 billion was spent for COPD care in the United States in 2010 and it is expected to be close to $50 billion in 2020.

Reducing healthcare utilization associated with COPD patient management (i.e. short-term readmission and chronic disease management) is a critically important unmet need for patients, caregivers, and hospitals. Early detection, prevention, and treatment of COPD exacerbation would aim to reduce this high morbidity and cost. To help reduce these exacerbations and improve disease management, sensors in a minimally invasive device can be used to identify factors that are associated with exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 45 years old
* Patient (or patient's legally authorized representative) is willing and able to provide written informed consent
* Patient is willing and able to comply with the protocol, including follow-up visits, electronic diary submissions and CareLink transmissions
* FEV1 (post bronchodilator) ≤ 70% of predicted
* Current or former smoker with lifetime cigarette consumption of > 10 pack-years
* One COPD exacerbation in the previous 12 months requiring hospitalization, urgent care or emergency department visit for respiratory illness OR Two COPD exacerbations within the previous 12 months requiring antibiotics and/or corticosteroids for respiratory symptoms.
* The patient's medical records must be accessible by the enrolling site over the follow-up period

Exclusion Criteria:

* Less than 30 days from diagnosis of a COPD exacerbation as defined as taking antibiotics and/or corticosteroids for respiratory symptoms, hospitalization, urgent care or emergency department visit for respiratory illness.
* Less than 30 days from diagnosis of a HF event as defined as any cardiovascular-related (including hypervolemia) Health Care Utilizations (HCUs) for any one of the following events:

  * Admission with primary diagnosis of HF
  * Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration at any one of the following settings:

    * Admission with secondary/tertiary diagnosis of HF
    * Emergency Department
    * Ambulance
    * Observation Unit
    * Urgent Care
    * HF/Cardiology Clinic
* Active respiratory infection being treated with antibiotics and/or corticosteroids
* Class IV heart failure
* Clinical diagnosis of unstable angina, bronchiectasis, or cystic fibrosis
* Any concomitant condition that might endanger the patient through participation in the study or interfere with study procedures, as assessed by the investigator
* Patient is pregnant (all females of child-bearing potential must have a negative pregnancy test within 1 week of enrollment)
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager
* Patient has an existing or planned implantation of Medtronic IPG, ICD, CRT-D or CRT-P device in the near future
* Patient has an existing and active insertable cardiac monitor, regardless of manufacturer
* Concurrent disease with life expectancy less than 1 year

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for the LINQ for COPD study is COPD patients who are known to have frequent exacerbations (one requiring hospitalization, ED visit, or urgent care visit, or at least two others in the past year).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Wendt, MD, Principal Investigator — U.S. Department of Veterans Affairs Minneapolis Healthcare System
Locations (9):
- United States (9):
  - Bay Area Cardiology Associates, Brandon, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Clinical Site Partners Inc, Leesburg, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Virtua Pulmonology Marlton, Marlton, New Jersey
  - Northwell Health Lenox Hill Hospital, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Lancaster General Hospital, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Though 42 subjects were enrolled, 2 subjects did not have successful Reveal LINQ insertions. Therefore, 40 subjects started the study.
Groups:
- Full Cohort: Participants had a successful Reveal LINQ insertion and investigational RAMware download.
Period: Overall Study
Arm/Group | Full Cohort
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Full Cohort
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40
Heart Rate [Mean (Standard Deviation); unit: bpm] — Baseline resting heart rate
  bpm | 80.5 (15.3)
Respiratory rate [Mean (Standard Deviation); unit: breaths per minute] — Baseline resting rate of respirations, breaths per minute Population: One subject was missing baseline respiratory rate measurement
  breaths per minute
    number analyzed (Participants) | 39
    (all) | 18.2 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: COPD Event
Description: Incidence of first COPD event
Time Frame: from subject randomization until 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 40
Participants | 28

ADVERSE EVENTS:
Time Frame: The data were collected from informed consent until death or study completion, two years
Description: All serious, LINQ system and procedure, pulmonary, and cardiovascular-related adverse events were collected throughout the study duration. The Endpoint Adjudication Committee reviewed all pulmonary-related AEs to determine COPD events.
Arm/Group | Full Cohort
All-Cause Mortality (participants affected / at risk) | 4/40
Serious Adverse Events (participants affected / at risk) | 27/40
Other Adverse Events (participants affected / at risk) | 24/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Cohort (N=40)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (8)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (4)
Death (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 1 (1)
Medical device site cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (8)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1)
Blood lactic acid increased (Investigations) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 (43)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Intermittent claudication (Vascular disorders) | 1 (2)
Shock (Vascular disorders) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Cohort (N=40)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Acute sinusitis (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 2 (3)
COVID-19 (Infections and infestations) | 4 (5)
Pneumonia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 18 (39)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04169529/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04169529/SAP_001.pdf